CLINICAL TRIAL: NCT02722070
Title: Processing Integration in Neurological Patients Using fMRI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0657-15-HMO-CTIL
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-01

CONDITIONS: Acute Inflammatory Demyelinating Polyradiculoneuropathy; Stroke; Anosognosia; Central and Peripheral Neurodegenerative Pathologies; Neuropsychiatric Conditions
MeSH Terms: conditions — Guillain-Barre Syndrome; Stroke; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy Controls: Age matched control for the various clinical groups
  Interventions: Device: 3 Tesla Siemens Skyra MRI scanner
- Neurodegenerative patients
  Interventions: Device: 3 Tesla Siemens Skyra MRI scanner
- Stroke patients
  Interventions: Device: 3 Tesla Siemens Skyra MRI scanner
- Neuropsychiatric patients
  Interventions: Device: 3 Tesla Siemens Skyra MRI scanner

INTERVENTIONS:
Device: 3 Tesla Siemens Skyra MRI scanner — Standardly used Magnetic resonance imaging (MRI) protocols, including resting state fMRI, task fMRI, T1 weighted imaging

SUMMARY:
The main objective of the study is to explore and map brain areas involved in processing and perception in patients suffering from neurological pathologies and condition. The investigators hypothesize for example, that a change (compare to healthy subjects) in the perceptual maps and body representation could be detected and characterize in patients suffering from impairments of peripheral nerve conduction.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of the investigated neuronal disease

Exclusion Criteria:

* contraindication for MRI scan
* pregnancy
* refusal to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffering from central and peripheral neurological pathologies and conditions
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-03; Primary Completion 2020-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic responses by measurement of the Blood-oxygen-level dependence(BOLD) signal | 2 years
  Distinct maps of sensory and multisensory representations related to certain disorders will be sassed by measurement of the Blood-oxygen-level dependence(BOLD) signal.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arzy S, Overney LS, Landis T, Blanke O. Neural mechanisms of embodiment: asomatognosia due to premotor cortex damage. Arch Neurol. 2006 Jul;63(7):1022-5. doi: 10.1001/archneur.63.7.1022. PMID 16831974